CLINICAL TRIAL: NCT06764017
Title: A Single-arm, Multicenter, Prospective Clinical Study of CHiR (chidamide, Zanubrutinib, and Lenalidomide) for Newly Diagnosed MYC- and BCL2-positive Diffuse Large B-cell Lymphoma (DLBCL) in Elderly Patients Intolerant to Chemotherapy.
Brief Title: CHiR Therapy for Elderly DLBCL Intolerant to Chemo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Lixia Sheng, Chief Physician, First Affiliated Hospital of Ningbo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-164A-02
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: diffuse large B-cell lymphoma; MYC- and BCL2-positive; chidamide; zanubrutinib; lenalidomide; elderly patients
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CHiR (Experimental): The combined regimen of chidamide, zanubrutinib, and lenalidomide (CHiR) is employed to treat elderly patients with double-expressor lymphoma. This study aims to explore the efficacy and safety of this regimen in newly diagnosed elderly patients with diffuse large B-cell lymphoma (DLBCL) who are intolerant to chemotherapy.
  Interventions: Drug: CHiR-DEL

INTERVENTIONS:
Drug: CHiR-DEL — Using the combined regimen of CHiR (chidamide, zanubrutinib, and lenalidomide) to treat newly diagnosed elderly patients with MYC- and BCL2-expressing positive diffuse large B-cell lymphoma (DLBCL) who are intolerant to chemotherapy.

SUMMARY:
The objective of exploring the application of CHiR is to evaluate its therapeutic efficacy and safety in newly diagnosed elderly patients with diffuse large B-cell lymphoma (DLBCL) aged 70 and above, and to investigate the genetic subtypes that may benefit from CHiR. The primary endpoint is the complete remission rate (CRR) at the end of 8 cycles.

ELIGIBILITY:
Inclusion Criteria：

1. Age ≥ 70 years;
2. ECOG score of 0-3;
3. Rated as unfit or frail on the simplified geriatric assessment (sGA);
4. Histologically confirmed CD20-positive diffuse large B-cell lymphoma (diagnostic criteria according to WHO 2016), excluding transformed type 2 DLBCL;
5. Immunohistochemically confirmed positive expression of MYC and BCL2 (MYC ≥ 40%, BCL2 ≥ 50% by immunohistochemistry);
6. Previously untreated patients;
7. Cardiac, hepatic, and renal function: creatinine < 2 times the upper limit of normal (ULN); ALT (alanine aminotransferase)/AST (aspartate aminotransferase) < 2.5 ULN; total bilirubin < 2 ULN;
8. At least one measurable lesion;
9. Unable to tolerate standard CHOP regimen chemotherapy or unwilling to receive chemotherapy;
10. Adequate understanding and voluntary signing of the informed consent form. Exclusion Criteria：

1.Patients with central nervous system involvement at the time of onset; 2.Known human immunodeficiency virus (HIV) infection; 3.Pregnant or lactating women; 4.Other tumors requiring treatment; 5.Uncontrollable active infection; 6.Active hepatitis with HBV-DNA copy number not controlled within 2*1000/mL despite antiviral treatment; 7.Inability to understand, comply with the study protocol, or sign the informed consent form.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
the complete remission rate (CRR) | Each cycle consists of 21 days, with a total of 8 cycles.
  The primary endpoint is the complete remission rate (CRR) at the end of 8 cycles.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No